CLINICAL TRIAL: NCT00394563
Title: A Randomized, Parallel Arm, Placebo-Controlled, Double-Blind, Multiple-Dose Study of the Safety and Efficacy of RN624 in Adults With Moderate-to-Severe Pain Due to Osteoarthritis of the Knee
Brief Title: A Phase II Study Looking at Moderate to Severe Osteoarthritis Knee Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trials Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091008; RN624-CL006
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis monoclonal antibody
MeSH Terms: conditions — Osteoarthritis | interventions — tanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): monoclonal antibody
  Interventions: Drug: RN624 (PF-04383119)
- 2 (Experimental)
  Interventions: Drug: RN624 (PF-04383119)
- 3 (Experimental)
  Interventions: Drug: RN624 (PF-04383119)
- 4 (Experimental)
  Interventions: Drug: RN624 (PF-04383119)
- 5 (Experimental)
  Interventions: Drug: RN624 (PF-04383119)
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: RN624 (PF-04383119) — 10 mcg/kg
  Arms: 1
Drug: RN624 (PF-04383119) — 25 mcg/kg
  Arms: 2
Drug: RN624 (PF-04383119) — 50 mcg/kg
  Arms: 3
Drug: RN624 (PF-04383119) — 100 mcg/kg
  Arms: 4
Drug: RN624 (PF-04383119) — 200 mcg/kg
  Arms: 5
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to look at the effects of RN624 on moderate to severe knee pain due to osteoarthritis. This study will look at the safety and pain relieving effects of RN624 compared to placebo over a 4 month period.

ELIGIBILITY:
Inclusion Criteria:

Male or non-pregnant female aged 40-75 with chronic moderate to severe knee pain due to OA (scoring 50 out of 100 on a visual analog scale on knee pain).

Subjects must meet one of the following: unwilling to take non-opiate pain medications, or for whom non-opiate pain medications have failed, or are candidates for or seeking invasive interventions such as intraarticular injections, knee arthroplasty, or total knee surgery

Exclusion Criteria:

History or symptoms of autoimmune disorders, cancer within the last 5 years except for cutaneous basal cell or squamous cell cancer resolved by excision, allergic reaction to monoclonal antibodies or IgG-fusion proteins, Hepatitis B, C or HIV, drug abuse, fibromyalgia, clinically significant cardiac disease, diabetes mellitus requiring oral treatment or insulin, clinically significant neurological disease or clinically significant psychiatric disorders

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Walking knee pain scores | Day 112

SECONDARY OUTCOMES:
Overall knee pain scores | Day 112
Incidence of adverse events and serious adverse events | Day 112
WOMAC | Day 112

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (45):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Cypress, California
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, Sacremento, California
  - Pfizer Investigational Site, Stamford, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Merrillville, Indiana
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Reno, Nevada
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Zanesville, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Midvale, Utah
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Yakima, Washington

REFERENCES:
- [Derived] Lane NE, Schnitzer TJ, Birbara CA, Mokhtarani M, Shelton DL, Smith MD, Brown MT. Tanezumab for the treatment of pain from osteoarthritis of the knee. N Engl J Med. 2010 Oct 14;363(16):1521-31. doi: 10.1056/NEJMoa0901510. Epub 2010 Sep 29. PMID 20942668
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091008&StudyName=A%20Phase%20II%20Study%20Looking%20at%20Moderate%20to%20Severe%20Osteoarthritis%20Knee%20Pain